CLINICAL TRIAL: NCT00437502
Title: A Phase I Study of Ovarian Cancer Peptides Plus GM-CSF and Adjuvant (Montanide ISA-51) as Consolidation Following Optimal Debulking and Systemic Chemotherapy for Women With Advanced Stage Ovarian, Tubal, or Peritoneal Cancer
Brief Title: A Phase I Study of Ovarian Cancer Peptides Plus GM-CSF and Adjuvant With Ovarian, Tubal or Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michael Morse, MD (Other)
Collaborators: Immunotope (Industry)
Responsible Party: Sponsor-Investigator, Michael Morse, MD, Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00013247; NCT00469677 (obsolete NCT alias)
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Epithelial Ovarian, Tubal or Peritoneal Cancer
Keywords: Immunotherapeutic vaccine; Ovarian cancer; epithelial ovarian cancer; tubal cancer; peritoneal cancer; immunotherapy
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- tumor peptide vaccine (Experimental): 2 cohorts: High and low dose tumor peptide vaccine
  Interventions: Biological: tumor peptide vaccine

INTERVENTIONS:
Biological: tumor peptide vaccine — Cohort 1 low dose level of vaccine @ 0.3 mg administered as x1 weekly injection given intradermally/subcutaneously into site assigned( same limb) for total number of study vaccine injections = 6.
Biological: tumor peptide vaccine — Cohort 2 high dose vaccine @ 1 mg administered as x1 weekly injection given intradermally/subcutaneously into site assigned( same limb) for total number of study vaccine injections = 6.

SUMMARY:
This study will evaluate the safety of administering a peptide vaccine consisting of twelve different tumor-rejection antigens known to be present on ovarian tumor cells. The vaccine is designed to elicit immune responses against twelve different pathways that are essential to tumor growth, survival and metastasis.HLA-A2+ is a required criteria for subject eligibility.

DETAILED DESCRIPTION:
The primary endpoint will be to determine the safety and feasibility of administering ovarian cancer peptides to women who have undergone debulking surgery and systemic chemotherapy, with the secondary objectives of evaluating immune response as measured by ELISPOT to the immunizations, to compare the immune response as measured by ELISPOT achieved by the two different dosing strategies and to assess disease relapse survival. Two cohorts of 9 patients each will be treated with different doses of the OCPM vaccine. They will receive the peptide vaccine subcutaneously on weeks 0,1,2,3,5 and6 and then receive the immunizations every 1 month for 6 months or disease recurrence. The first 9 patients will be entered into the first cohort; if 1 or fewer patients experience Dose-limiting toxicity (DLT) then the next 9 will be enrolled into the second cohort. DLT is defined as any Grade 3 or greater hematologic or non-hematologic toxicity or autoimmune disease (except for fever, skin reaction, or alopecia which would be grade 4) occurring at any time from the first immunization until 30 days after the last immunization. Toxicity will be assessed at each dose level using CTC toxicity criteria. Ovarian cancer peptide-specific immune response will be measured by ELISpot. Time to disease relapse will be based on composite assessment of clinical signs, objective exam findings, radiologic imaging, and CA125 results. A dosing scheme will be considered safe if <1 of the first 9 subjects treated at a dose level experience DLT (as described above). A subject will be considered evaluable for safety if treated with at least one immunization. A T cell response will be considered positive by ELISpot if: the mean number of spots in six wells with antigen exceeds the number of spots in six control wells by 10 and the difference between single values of the six wells containing antigen and the six control wells is statistically significant at a level of p ≤ 0.05 using Student's t test.

ELIGIBILITY:
Inclusion Criteria:

Must be HLA-A2+ patients with histologically confirmed, stage III-IV epithelial ovarian, tubal, or peritoneal cancer who have undergone optimal debulking and had a complete clinical response to front-line platin/taxane based chemotherapy.

* Subjects must have received front-line platin compound and taxane chemotherapy following primary surgical resection. Front-line treatment can include up to 12 cycles of treatment.Subjects must receive the first dose of study medication at least 4 weeks and up to 6 months since completing their last dose of front-line chemotherapy.A complete clinical response defined as: no evidence of disease on physical exam,CT imaging scans of the abdomen and pelvis, chest x-ray and a CA-125 below the upper limit of normal.

Exclusion Criteria:

* History of autoimmune disease, serious intercurrent chronic or acute illness, active hepatitis, serologic evidence for HIV, splenectomy, or be receiving steroid or immunosuppressive therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Date of first objective finding will be used to define the date of relapse | From date of enrollment to date of confirmed relaspe

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morse, MD, Principal Investigator — Duke University; Angeles A Secord, MD, Principal Investigator — Duke University; Ramila Philip, PhD, Principal Investigator — Immunotope
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Morse MA, Secord AA, Blackwell K, Hobeika AC, Sinnathamby G, Osada T, Hafner J, Philip M, Clay TM, Lyerly HK, Philip R. MHC class I-presented tumor antigens identified in ovarian cancer by immunoproteomic analysis are targets for T-cell responses against breast and ovarian cancer. Clin Cancer Res. 2011 May 15;17(10):3408-19. doi: 10.1158/1078-0432.CCR-10-2614. Epub 2011 Feb 7. PMID 21300761